CLINICAL TRIAL: NCT04648579
Title: Automated Documentation of Vital Parameters in Wards Using Mobile Stations - Effect on the Appropriate Activation of the Rapid Response Team: a Cluster Randomized Clinical Trial
Brief Title: Automated Documentation of Vital Parameters Using Mobile Stations and Activation of the Rapid Response Team
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital do Coracao (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HILLROM
Record Dates: First submitted 2020-11-23; First posted 2020-12-01 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2022-02

CONDITIONS: Inpatient Facililty Diagnoses

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hillrom (Experimental): The intervention involves an automated vital signs document system consisting of a mobile medical device for measuring vital signs (CSM / Hillrom) that collects and analyzes data acquired at the bedside to be sent to a remote data processing point (Digital Control Station), using Hillrom Connecta software.
  Interventions: Device: Hillrom
- Control (Active Comparator): Hospital usual care.
  Interventions: Other: Control

INTERVENTIONS:
Device: Hillrom — Hillrom Connecta solution will record vital signs in an automated way, without the need for human intervention, and activate TRR activation when at least one criteria is met. The frequency of monitoring vital signs will be defined based on the MEWS score.
  Arms: Hillrom
Other: Control — Hospital usual care regarding vital signs collection and TRR activation.
  Arms: Control

SUMMARY:
The documentation of vital signs is traditionally performed manually when the patient is not admitted in intensive care units, which can lead to documentary errors, long time for data acquisition and, consequently, impairment in the early identification of possible clinical deterioration. In-bed technology solutions are available to automate the collection of vital data and transfer information to a medical record or central electronic monitoring and its role in the health value chain needs further investigation. The investigators propose to evaluate the impact of the Connex Spot Monitor solution Welch Allyn (CSM / Hillrom) in conjunction with the Hillrom Connecta solution in a real world situation, conducting a cluster randomized trilal in wards of a tertiary hospital. In addition, this study aims to estimate the clinical effectiveness of a technological solution that performs an analysis of vital signs and automatically activates the rapid response team (RRT) when the pre-defined criteria are met, comparing it with the traditional manual method. The primary outcome is the number of times that the RRT fires in a timely manner.

ELIGIBILITY:
Inclusion Criteria:

- All patients with activated RRT during the study recruitment period.

Exclusion Criteria:

- Individuals who need blood pressure measurement in lower members.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 231 (Actual)
Dates: Start 2021-04-22 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
RRT | 24 hours
  Number of rapid response team triggers activated in a timely manner.

CONTACTS AND LOCATIONS:
Overall Officials: José César Ribeiro, RN, Principal Investigator — Hospital do Coracao
Locations (1):
- Hospital do Coracao, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data will be available upon reasonable request including a short study protocol. Both sponsor and funders will evaluate all requests. Brazilian regulatory agencies approval will be also required.
Supporting Information: Study Protocol
Time Frame: After main paper publication.

REFERENCES:
- [Derived] Ribeiro JC, Sgorbissa C, Silva KA, Braz MLD, Horak ACP, Nicola ML, Gurgel RM, Tokunaga SM, Negrelli KL, Murizine GS, Medrado Junior F, Coli RCP, Cavalcanti AB, Marcadenti A. Automated documentation of vital parameters in wards using portable stations - Effect on proper triggering of the rapid response team: a study protocol of a cluster randomized clinical trial. Rev Bras Ter Intensiva. 2022 Nov 4;34(3):319-326. doi: 10.5935/0103-507X.20220101-pt. eCollection 2022. PMID 36351064